CLINICAL TRIAL: NCT03847571
Title: Acetazolamide (AZ) for Management of Refractory Hypokalemia Metabolic Alkalosis in Bartter Syndrome
Brief Title: Acetazolamide (AZ) for Management of Alkalosis in Bartter Syndrome
Acronym: AZ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: Acetazolamide (AZ)
Record Dates: First submitted 2019-02-16; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Bartter Syndrome
Keywords: Acetazolamide; Hypokalemic metabolic alkalosis; Bartter syndrome
MeSH Terms: conditions — Bartter Syndrome | interventions — Acetazolamide

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acetazolamide: Oral administration of acetazolamide 5 mg/kg/day for 4 weeks
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Acetazolamide — Correction of metabolic alkalosis by inhibition of the filtered bicarbonate load reabsorption in the proximal tubules using acetazolamide (AZ)

SUMMARY:
In this prospective controlled cross over clinical trial, the investigators aim to evaluate the efficacy and safety of acetazolamide for the management of metabolic alkalosis in children with Bartter syndrome. Urine and blood electrolytes will be measured before and after acetazolamide treatment. The primary end point is a change in polyuria, hypokalemia, and metabolic alkalosis.

DETAILED DESCRIPTION:
Bartter syndrome is a hereditary salt-loosing tubulopathy caused by several gene mutations encoding the sodium reabsorption in the thick ascending limb of loop of Henle, with poor response to treatment. The effects of inhibition of proximal tubular reabsorption of bicarbonate by acetazolamide have not been previously studied in Batter patients.

The present study is designed to assess he efficacy and safety of acetazolamide for the management of children with Bartter syndrome. The primary end point is change in polyuria, hypokalemia, and metabolic alkalosis.

In this prospective observational crossover clinical trial, patients between ages 1 and 10 years with clinical diagnosis of Bartter syndrome (hypokalemia, metabolic alkalosis, normal blood pressure, elevated urine chloride >20 milliequivalent per liter, high serum aldosterone and plasma renin levels) will be enrolled in a 4- week clinical trial. After initial clinical and laboratory evaluations, patients will receive acetazolamide 5.0 mg/kg orally as a single daily dose and each patient will act as his/her own control. Renal electrolyte and 24-hour urine output will be measured at baseline and after the 4 weeks acetazolamide treatment.

ELIGIBILITY:
Inclusion Criteria:

* Hypokalemia
* metabolic alkalosis
* normal blood pressure
* random urine chloride >20 milliequivalent per liter (mEq/L)
* Elevated serum aldosterone and renin levels

Exclusion Criteria:

* Hypertension
* History of emesis
* Prior use of laxatives
* Cystic fibrosis ofpancrease

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between 1 and 10 years of age with failure to thrive, polyuria and unexplained hypokalemic metabolic alkalosis will be recruited for this trial.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Metabolic alkalosis | 4 weeks
  Change in serum bicarbonate level
Urine output | 4 weeks
  Change in 24-hr urine volume

CONTACTS AND LOCATIONS:
Overall Officials: Farahnak Assadi, MD, Study Director — Rush University Medical Center
Locations (4):
- Iran (4):
  - Fateme Ghane Sharbaf, Mashhad
  - Semnan University of Medical Sciences, Semnan
  - Banafshe Dormansh, Tehran
  - Simin Sadeghi, Zahedan